CLINICAL TRIAL: NCT00437853
Title: Neoadjuvant Hormonal Treatment of Postmenopausal Women Who Have Operable Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cancerologia de Mexico (Other)
Collaborators: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1033MX/0001; NCT00262535 (obsolete NCT alias)
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2007-02-21 (Estimated); Status verified 2007-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

INTERVENTIONS:
Drug: Anastrozole

SUMMARY:
EFFICACY OF NEOADJUVANT ENDOCRINE THERAPY WITH ANASTROZOLE IN POMENOPAUSAL WOMEN WITH ER-POSITIVE BREAST CANCER.

Flavia Morales-Vásquez, Horacio Noé López Basave.

Background: Neoadjuvant Hormonal Therapy (HT) is being used increasingly to downstage locally advanced and large operable breast cancer. Following this treatment, inoperable breast cancer often becomes fully respectable and tumors requiring mastectomy may be successfully removed by breast-conserving surgery (BCS).

Methods: Recruit postmenopausal women with ER(+) and/or PgR (+) breast cancer (BC) T2,N1-2 to T3,N0-1 were assigned to HT with anastrozole 1 mgr daily for 4 months.

The primary endpoint was to compare overall objective response (OR) determined by clinical (palpation) and ultrasound. Secondary endpoint was the number of patients who qualified for BCS plus radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women who had primary breast cancer, histological confirmed, through a core needle biopsy, and who{s tumors positive for estrogens receptor ER/PR.

Clinical stage IIB or IIIA Tumor assessable by clinical exam, mammogram or and ultrasound Adequate functional bone marrow Documented evidence adequate renal function and liver function Life expectancy for six months Written inform consent

Exclusion Criteria:

* Prior treatment with letrozole or tamoxifen uncontrol disorders patients with instable angina or uncontrol cardiac disease patient with bilateral breast tumors patients elegies for conservative breast surgery Inflammatory breast cancer o distant metastases Other concurrent malignancies, except carcinoma with in situ cono biopsy of uterine cervix or adequate treat skin cancer no melanoma concomitant cancer treatment such as chemotherapy, immunotherapy biological modulators, endocrinotherapy, biphosphonates therapy and radiotherapy.

Concomitant treatment with steroids Others research drug whiting the last 30 days and concomitant use of research drugs History non compliance with medications schedules and patients consider potential unreliable.

Min Age: 66 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30
Dates: Start 2003-06; Study Completion 2007-02

PRIMARY OUTCOMES:
The primary endpoint was to compare overall objective response (OR) determined by clinical (palpation) and ultrasound.

SECONDARY OUTCOMES:
Secondary endpoint was the number of patients who qualified for BCS plus radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Morales-Vasquez, Principal Investigator — Instituto Nacional de Cancerologia Mexico; Alejandro Mohar, Study Director — Instituto Nacional de Cancerologia Mexico; Alfonso Dueñas Gonzalez, Study Chair — Instituto Nacional de Cancerologia de Mexico
Locations (1):
- Instituto Nacional de Cancerologia de Mexico, Mexico City, Mexico City, Mexico